CLINICAL TRIAL: NCT03356756
Title: Diagnostic and Prognostic Significance of Combined PET/MRI in Inflammatory Cardiomyopathies and Sarcoidosis
Brief Title: PET MRI Study in Patients With Cardiac Sarcoidosis
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 15-9933
Record Dates: First submitted 2017-11-03; First posted 2017-11-29 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Cardiomyopathy; Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PET MRI exam: simultaneous combined 18F-FDG PET and cardiac MRI imaging (PET MRI) performed immediately after the PET CT exam.
  Interventions: Diagnostic Test: simultaneous combined 18F-FDG PET and cardiac MRI imaging

INTERVENTIONS:
Diagnostic Test: simultaneous combined 18F-FDG PET and cardiac MRI imaging — Patients will undergo a research study performed with an integrated whole-body PET/MRI imaging system designed for simultaneous PET and MRI acquisition, immediately after standard of care PET/CT exam.

SUMMARY:
Myocarditis or inflammatory cardiomyopathy refers to inflammation of the heart muscle (the myocardium). Sarcoidosis is a multisystem granulomatous disorder that may involve the heart, causing inflammation, and potentially resulting in complications including arrhythmia and sudden death. The objective of this study is to evaluate the diagnostic and prognostic significance of simultaneous combined 18F-FDG PET and cardiac MRI imaging in the evaluation of inflammatory cardiomyopathies including cardiac sarcoidosis. Combined PET/MRI imaging may allow for detection and quantification of active myocardial inflammation as well as chronic fibrosis and scarring. Results of this study may allow for earlier detection of cardiac inflammation when compared with methods in current clinical use, and may lead to better understanding of the disease processes contributing to adverse outcomes. Elucidation of imaging findings associated with future adverse event risk may impact patient management such as providing an indication for pacemaker or defibrillator implantation, or escalation of medical therapy.

DETAILED DESCRIPTION:
Myocarditis or inflammatory cardiomyopathy refers to inflammation of the myocardium. Sarcoidosis is a multisystem granulomatous disorder of unknown etiology, which can result in myocardial inflammation. Approximately 5% of patients with sarcoidosis have clinically apparent cardiac involvement, yet autopsy series indicate that cardiac involvement is present in up to 25% of cases. This discrepancy suggests that cardiac sarcoidosis may be under-diagnosed in clinical practice. Recent studies have demonstrated high diagnostic accuracy of both cardiac MRI and 18F-labelled fluoro-2-deoxyglucose (FDG) PET for detection of cardiac involvement. However, cardiac MRI may fail to identify areas of active inflammation even with fluid sensitive T2-weighted sequences.

Fasting 18F-FDG positron emission tomography (PET) has been shown to identify early cardiac sarcoidosis with relatively high sensitivity. To date, simultaneous PET/MRI evaluation of cardiac inflammation and sarcoidosis has only been described in limited case reports. The objective of the proposed research is to evaluate the utility of simultaneous PET/MRI imaging in patients with cardiac sarcoidosis and other inflammatory cardiomyopathies.

ELIGIBILITY:
Inclusion Criteria:

* The primary criterion for enrolment will be patients ≥18 years of age with known or suspected sarcoidosis or other inflammatory cardiomyopathy who are referred for clinically indicated 18F-FDG PET/CT imaging

Exclusion Criteria:

* Standard cardiac MRI contraindications include arrhythmia, claustrophobia, history of allergic reaction or other contraindication to gadolinium-based contrast agent, impaired renal function with eGFR < 60 ml/min/1.73m2, pregnancy, breast-feeding, or any other general contraindication to MRI (pacemaker, cerebral aneurysm clips, shrapnel, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with known or suspected cardiac sarcoidosis or other inflammatory cardiomyopathy who are referred for clinically indicated 18F-FDG PET/CT imaging at University Health Network.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
The incremental value of combined 18F-FDG PET and cardiac MRI imaging in the evaluation of patients with suspected cardiac sarcoidosis or cardiac inflammation | Completion of enrollment, an average of two years
  Patients will undergo standard clinical evaluation using modified consensus guidelines for the diagnosis of sarcoidosis. Following enrolment, patients will also undergo parallel assessment for cardiac involvement by PET/MRI. Comparison of cardiac involvement identified by modified consensus criteria and PET/MRI will be performed.

SECONDARY OUTCOMES:
The differences in circulating plasma biomarkers between cardiac with suspected cardiac sarcoidosis and healthy people | Completion of enrollment, an average of two years
  A cohort of 25 healthy volunteers will be recruited for comparison of patients with suspected cardiac sarcoidosis. Biomarkers such as microRNA will be analyzed in both groups.
The prognostic significance of PET-MRI imaging findings in patients with cardiac inflammation | Through study completion, an average of three years
  Clinical follow-up to track adverse events to validate imaging findings and determine their prognostic significance.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hanneman, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Result] Cheung E, Ahmad S, Aitken M, Chan R, Iwanochko RM, Balter M, Metser U, Veit-Haibach P, Billia F, Moayedi Y, Ross HJ, Hanneman K. Combined simultaneous FDG-PET/MRI with T1 and T2 mapping as an imaging biomarker for the diagnosis and prognosis of suspected cardiac sarcoidosis. Eur J Hybrid Imaging. 2021 Dec 16;5(1):24. doi: 10.1186/s41824-021-00119-w. PMID 34913098
- [Result] Marschner CA, Aloufi F, Aitken M, Cheung E, Thavendiranathan P, Iwanochko RM, Balter M, Moayedi Y, Duero Posada J, Hanneman K. Combined FDG PET/MRI versus Standard-of-Care Imaging in the Evaluation of Cardiac Sarcoidosis. Radiol Cardiothorac Imaging. 2023 Sep 28;5(5):e220292. doi: 10.1148/ryct.220292. eCollection 2023 Oct. PMID 38076597